CLINICAL TRIAL: NCT03436940
Title: Comparison Between Two Strategies of Discharge Planning for the Reduction of Short Term Hospital Readmissions: A Cluster Randomized Cross-over Trial
Brief Title: Comparison Between Two Strategies of Discharge Planning for the Reduction of Short Term Hospital Readmissions
Acronym: PROMENADE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Principal Investigator, Daniela Corsi, MD, Director of "SSD Integrazione Ospedale-Territorio", A.O.U. Città della Salute e della Scienza
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CS2/378/2017
Record Dates: First submitted 2018-02-13; First posted 2018-02-19 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Patient Discharge

STUDY DESIGN:
Intervention Model Description: cluster randomized cross-over trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- On Demand Discharge Planning (DDP) (Active Comparator): Patients with an intermediate score, according to the simplified Blaylock Risk Assessment Screening Score, are addressed to the NOCC team only in case of a specific request by the unit of hospitalization.
  Interventions: Other: On Demand Discharge Planning (DDP)
- Routine Discharge Planning (RDP) (Experimental): All patients with an intermediate threshold value of the simplified Blaylock Risk Assessment Screening Score are submitted to discharge planning by the NOCC team (Hospital Unit of Continuity of Care)
  Interventions: Other: Routine Discharge Planning (RDP)

INTERVENTIONS:
Other: On Demand Discharge Planning (DDP) — Patients with an intermediate score, according to the simplified Blaylock Risk Assessment Screening Score, are addressed to the NOCC team (hospital Continuity of care team) only in case of a specific request by the unit of hospitalization.
  Arms: On Demand Discharge Planning (DDP)
Other: Routine Discharge Planning (RDP) — All patients with an intermediate threshold value of the simplified Blaylock Risk Assessment Screening Score are submitted to discharge planning by the NOCC team (Hospital Unit of Continuity of Care)
  Arms: Routine Discharge Planning (RDP)

SUMMARY:
The purpose of this study is to improve discharge planning effectiveness by comparing two strategies [on-Demand Discharge Planning (DDP) vs. Routine Discharge Planning (RDP)], in terms of reduction of hospital readmissions for inpatients classified at intermediate risk of complex discharge using the simplified Blaylock Risk Assessment Screening Score (BRASS).

DETAILED DESCRIPTION:
The purpose of this study is to improve discharge planning effectiveness by comparing two strategies [on-Demand Discharge Planning (DDP) vs. Routine Discharge Planning (RDP)], in terms of reduction of hospital readmissions for inpatients classified at intermediate risk of complex discharge using the simplified Blaylock Risk Assessment Screening Score (BRASS).

Five Internal Medicine Unit and four Units of Neurology will be randomized to the two different strategies of discharge planning (RDP or DDP), based on two different alternating sequences of four periods (each period comprising three months). The randomization will be stratified by type of unit.

Patients at risk of complex discharge, according to the simplified BRASS score, are assigned to the Hospital Unit of Continuity of Care (NOCC) team, using the hospital telematics system. Afterwards, the NOCC team proposes an appropriate discharge planning, considering clinical and social needs.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients (age ≥ 18 years);
* Residents in Piedmont, Italy;
* Patients admitted to General Internal Medicine or Neurology Units of Molinette Hospital (Turin)
* Patients with a score in the simplified BRASS between 4 and 6 at admission

No specific exclusion criteria were applied.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 802 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-10-12 (Actual); Study Completion 2019-10-13 (Actual)

PRIMARY OUTCOMES:
Unexpected hospital readmission within 90 days from discharge | 90 days
  Proportion of hospital admissions in the standard admission regime within 90 days from the date of discharge. The endpoint will be calculated only for patients discharged alive. Readmissions for any cause under ordinary admissions will be considered as event. The Day Hospital re-admissions will not be considered for the endpoint calculation.

SECONDARY OUTCOMES:
Proportion of Long Length of Stay (LLOS) | 150 days
  Proportion of admissions with long duration of hospitalization (LLOS - Long Length of Stay). The endpoint will be calculated for all hospitalized patients. An admission will be considered as LLOS if its duration will be higher than the 90th specific percentile for Diagnostic Related Group (DRG ) detected at the regional level in Piedmont in 2016.
Death within 90 days from discharge | 90 days
  Proportion of deaths within 90 days of discharge date. The endpoint will be calculated only for patients discharged alive. Death for any cause will be considered as event.
Proportion of patients reported to the NOCC team during the DDP-experimental phase | 150 days
  Incidence of activations of the NOCC in the periods of adoption of the DDP strategy (only for admissions treated with DDP strategy)
Healthcare costs until 90 days from the discharge | 90 days
  Health care costs charged to the National Health Service (NHS) between the date of admission and 90 days from the date of discharge or death of the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Corsi, MD, Principal Investigator — A.O.U. Città della Salute e della Scienza
Locations (1):
- AOU Città della Salute, Torino, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Evangelista A, Camussi E, Corezzi M, Gilardetti M, Fonte G, Scarmozzino A, La Valle G, Angelone L, Olivero E, Ciccone G, Corsi D. Routine vs. On-Demand Discharge Planning Strategy in Intermediate-Risk Patients for Complex Discharge: a Cluster-Randomized, Multiple Crossover Trial. J Gen Intern Med. 2023 Sep;38(12):2749-2754. doi: 10.1007/s11606-023-08186-4. Epub 2023 May 11. PMID 37170018